CLINICAL TRIAL: NCT03770182
Title: Brain Stimulation for Neurological Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Storz Medical AG (Industry)
Collaborators: Medical University of Vienna (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TPS-AD-Vienna
Record Dates: First submitted 2018-09-07; First posted 2018-12-10 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): NEUROLITH
  * Cycle 1: Active treatment
  * Cycle 2: Sham treatment
  Interventions: Device: NEUROLITH
- Group B (Experimental): NEUROLITH
  * Cycle 1: Sham treatment
  * Cycle 2: Active treatment
  Interventions: Device: NEUROLITH

INTERVENTIONS:
Device: NEUROLITH — transcranial pulse stimulation (TPS)
  Other Names: transcranial pulse stimulation; TPS

SUMMARY:
This is a prospective double-blind randomized placebo-controlled crossover clinical trial

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable patients with probable Alzheimer's Disease (Diagnosis according to ICD-10 Criteria (F00))
* At least 3 months of stable antidementive therapy or no antidementive therapy necessary
* Signed written informed consent
* Monthly pregnancy test for women in childbearing years
* Age >= 18 years

Exclusion Criteria:

* Non-compliance with the protocol
* Pregnant or breastfeeding women
* Relevant intracerebral pathology unrelated to the Alzheimers's disease (e.g. Brain tumor)
* Hemophilia or other blood clotting disorders
* Cortisone treatment within the last 6 weeks before first treatment
* Thrombosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
Consortium to Establish a Registry for Alzheimer's Disease (CERAD) - Corrected Total Score | month 3
  CERAD stands for "The Consortium to Establish a Registry for Alzheimer's Disease". The CERAD was funded by the National Institute on Aging in 1986 to develop standardized, validated measures for the assessment of Alzheimer's disease (Fillenbaum 2008). CERAD is a cognitive test battery which is normalized for age, gender and education (Morris 1988). The CERAD total score (Chandler 2005) is a good measure for Alzheimer's Disease (Ehrensperger 2010, Rossetti 2010, Seo 2010, Hallikainen 2013).
  The CERAD total score is a scale from 0 to 100 with 100 meaning "normal cognitive ability" and 0 meaning "severe cognitive impairment".

SECONDARY OUTCOMES:
Alzheimer's Disease Assessment Scale (ADAS) | immediately post-treatment
  Cognitive test. The Alzheimer's Disease Assessment Scale (ADAS) was designed to evaluate the severity of cognitive and noncognitive behavioral dysfunctions characteristic of persons with Alzheimer's disease (Rosen 1984). It consists of 21 items. Its sensitivity seems limited in mild AD (Irizarry 2008) but it is commonly used with AD intervention studies.
  The ADAS total score (ADASUM) ranges from 0 to 120 and consists of two subscales, the ADAS-COG with 70 possible points and the ADAS-NonCog with 50 possible points. In both subscales and total scale 0 points means "healthy" and the highest score means "severe impairment". The total score ADASUM is the sum of both subscales.
  Its cognition subscale (ADAS-COG) is a standard tool in pivotal clinical trials to detect therapeutic efficacy in cognition (Robert 2010). The ADAS-COG includes 11 items assessing the several cognitive domains.
Alzheimer's Disease Assessment Scale (ADAS) | month 1
  Cognitive test. The Alzheimer's Disease Assessment Scale (ADAS) was designed to evaluate the severity of cognitive and noncognitive behavioral dysfunctions characteristic of persons with Alzheimer's disease (Rosen 1984). It consists of 21 items. Its sensitivity seems limited in mild AD (Irizarry 2008) but it is commonly used with AD intervention studies.
  The ADAS total score (ADASUM) ranges from 0 to 120 and consists of two subscales, the ADAS-COG with 70 possible points and the ADAS-NonCog with 50 possible points. In both subscales and total scale 0 points means "healthy" and the highest score means "severe impairment". The total score ADASUM is the sum of both subscales.
  Its cognition subscale (ADAS-COG) is a standard tool in pivotal clinical trials to detect therapeutic efficacy in cognition (Robert 2010). The ADAS-COG includes 11 items assessing the several cognitive domains.
Alzheimer's Disease Assessment Scale (ADAS) | month 3
  Cognitive test. The Alzheimer's Disease Assessment Scale (ADAS) was designed to evaluate the severity of cognitive and noncognitive behavioral dysfunctions characteristic of persons with Alzheimer's disease (Rosen 1984). It consists of 21 items. Its sensitivity seems limited in mild AD (Irizarry 2008) but it is commonly used with AD intervention studies.
  The ADAS total score (ADASUM) ranges from 0 to 120 and consists of two subscales, the ADAS-COG with 70 possible points and the ADAS-NonCog with 50 possible points. In both subscales and total scale 0 points means "healthy" and the highest score means "severe impairment". The total score ADASUM is the sum of both subscales.
  Its cognition subscale (ADAS-COG) is a standard tool in pivotal clinical trials to detect therapeutic efficacy in cognition (Robert 2010). The ADAS-COG includes 11 items assessing the several cognitive domains.
Neuropsychological Test Battery Vienna (NTBV) | immediately post-treatment
  The Neuropsychological Test Battery Vienna (NTBV) ist a cognitive test, which was created to detect Alzheimer's Disease (Lehrner 2007).
Neuropsychological Test Battery Vienna (NTBV) | month 1
  Cognitive test
Neuropsychological Test Battery Vienna (NTBV) | month 3
  Cognitive test
CERAD | immediately post-treatment
  Cognitive test
CERAD | month 1
  Cognitive test
CERAD | month 3
  Cognitive test
Clock drawing test | immediately post-treatment
  The clock drawing test shows the visuoconstructive skills (Shulman 1986). The subject is asked to draw the face of a clock with all numbers and to set the hands for a specified time (hh:mm). Scores range from 0 (worst) to 7 (best).
Clock drawing test | month 1
  Clock drawing test
Clock drawing test | month 3
  Clock drawing test
Forgetfulness assessment inventory (FAI) | immediately post-treatment
  FAI stands for "Forgetfulness Assessment Inventory". The Forgetfulness Assessment Inventory is a questionnaire. Kogler et al (2013) developed the forgetfulness assessment inventory FAI (German: Skala zur Erfassung der Gedächtnisleistung - SEG) to evaluate subjective complaints regarding everyday memory problems. Lehrner et al. (2014) validated the test. The FAI consists of 16 items to measure subjective memory problems in daily life based on a Likert scale.
  The FAI focuses on the subjective evaluation of memory problems, particularly in relation to episodic memory, which has been found to be very sensitive in the early detection of mild cognitive impairment and AD (Lehrner 2014). This questionnaire is supposed to be completed by the patient as well as by a person familiar with the patient.
  The total score ranges from 0 to 80. Higher scores reflect poorer subjective functioning and greater complaints.
Forgetfulness assessment inventory (FAI) | month 1
  FAI stands for "Forgetfulness Assessment Inventory". The Forgetfulness Assessment Inventory is a questionnaire. Kogler et al (2013) developed the forgetfulness assessment inventory FAI (German: Skala zur Erfassung der Gedächtnisleistung - SEG) to evaluate subjective complaints regarding everyday memory problems. Lehrner et al. (2014) validated the test. The FAI consists of 16 items to measure subjective memory problems in daily life based on a Likert scale.
  The FAI focuses on the subjective evaluation of memory problems, particularly in relation to episodic memory, which has been found to be very sensitive in the early detection of mild cognitive impairment and AD (Lehrner 2014). This questionnaire is supposed to be completed by the patient as well as by a person familiar with the patient.
  The total score ranges from 0 to 80. Higher scores reflect poorer subjective functioning and greater complaints.
Forgetfulness assessment inventory (FAI) | month 3
  FAI stands for "Forgetfulness Assessment Inventory". The Forgetfulness Assessment Inventory is a questionnaire. Kogler et al (2013) developed the forgetfulness assessment inventory FAI (German: Skala zur Erfassung der Gedächtnisleistung - SEG) to evaluate subjective complaints regarding everyday memory problems. Lehrner et al. (2014) validated the test. The FAI consists of 16 items to measure subjective memory problems in daily life based on a Likert scale.
  The FAI focuses on the subjective evaluation of memory problems, particularly in relation to episodic memory, which has been found to be very sensitive in the early detection of mild cognitive impairment and AD (Lehrner 2014). This questionnaire is supposed to be completed by the patient as well as by a person familiar with the patient.
  The total score ranges from 0 to 80. Higher scores reflect poorer subjective functioning and greater complaints.
Instrumental Activities of Daily Living Scale (IADL) - Patient | immediately post-treatment
  IADL stands for "Instrumental Activities of Daily Living". Lawton's Instrumental Activities of Daily Living Scale (IADL) is an instrument to assess independent living skills (Lawton 1969). This questionnaire is supposed to be completed by the patient as well as by a person familiar with the patient. There are 8 domains of function measured with the Lawton IADL scale: Telephone, Shopping, Food preparation, Housekeeping, Laundry, Mode of transportation, Medication, Finances.
  The Total Score is a sum of all domains. The total score ranges from 0 (low function, dependent) to 8 (high function, independent). For male patients the highest possible score is 5 (due to expected zero scores for food preparation, housekeeping, and laundry).
IADL- Patient | month 1
  IADL stands for "Instrumental Activities of Daily Living". Lawton's Instrumental Activities of Daily Living Scale (IADL) is an instrument to assess independent living skills (Lawton 1969). This questionnaire is supposed to be completed by the patient as well as by a person familiar with the patient. There are 8 domains of function measured with the Lawton IADL scale: Telephone, Shopping, Food preparation, Housekeeping, Laundry, Mode of transportation, Medication, Finances.
  The Total Score is a sum of all domains. The total score ranges from 0 (low function, dependent) to 8 (high function, independent). For male patients the highest possible score is 5 (due to expected zero scores for food preparation, housekeeping, and laundry).
IADL- Patient | month 3
  IADL stands for "Instrumental Activities of Daily Living". Lawton's Instrumental Activities of Daily Living Scale (IADL) is an instrument to assess independent living skills (Lawton 1969). This questionnaire is supposed to be completed by the patient as well as by a person familiar with the patient. There are 8 domains of function measured with the Lawton IADL scale: Telephone, Shopping, Food preparation, Housekeeping, Laundry, Mode of transportation, Medication, Finances.
  The Total Score is a sum of all domains. The total score ranges from 0 (low function, dependent) to 8 (high function, independent). For male patients the highest possible score is 5 (due to expected zero scores for food preparation, housekeeping, and laundry).
Beck Depression Inventory (BDI) | immediately post-treatment
  BDI stands for the "Beck Depression Inventory". The Beck Depression Inventory (BDI) measures the severity of depression (Beck 1961). It is a 21-item questionnaire for self-evaluation with 0-3 scores per item. The total score is the sum of all items. It ranges from 0 (normal state) to 63 (severe depression).
Beck Depression Inventory (BDI) | month 1
  BDI stands for the "Beck Depression Inventory". The Beck Depression Inventory (BDI) measures the severity of depression (Beck 1961). It is a 21-item questionnaire for self-evaluation with 0-3 scores per item. The total score is the sum of all items. It ranges from 0 (normal state) to 63 (severe depression).
Beck Depression Inventory (BDI) | month 3
  BDI stands for the "Beck Depression Inventory". The Beck Depression Inventory (BDI) measures the severity of depression (Beck 1961). It is a 21-item questionnaire for self-evaluation with 0-3 scores per item. The total score is the sum of all items. It ranges from 0 (normal state) to 63 (severe depression).
Prosopagnosia index (PI20) | immediately post-treatment
  PI20 stands for the "20-item prosopagnosia index". The PI20 is a self-report instrument for identifying developmental prosopagnosia, also called face blindness. Patients indicate the extent to which 20 statements describe their face recognition experiences. Each statement is scored on a five-point scale. The total score is the sum of all scores. It ranges from 0 to 100. Higher scores reflect impairment to recognize faces.
Prosopagnosia index (PI20) | month 1
  PI20 stands for the "20-item prosopagnosia index". The PI20 is a self-report instrument for identifying developmental prosopagnosia, also called face blindness. Patients indicate the extent to which 20 statements describe their face recognition experiences. Each statement is scored on a five-point scale. The total score is the sum of all scores. It ranges from 0 to 100. Higher scores reflect impairment to recognize faces.
Prosopagnosia index (PI20) | month 3
  PI20 stands for the "20-item prosopagnosia index". The PI20 is a self-report instrument for identifying developmental prosopagnosia, also called face blindness. Patients indicate the extent to which 20 statements describe their face recognition experiences. Each statement is scored on a five-point scale. The total score is the sum of all scores. It ranges from 0 to 100. Higher scores reflect impairment to recognize faces.
Neuropsychiatric Inventory (NPI) (Care Taker) | immediately post-treatment
  The NPI stands for "Neuropsychiatric Inventory". It is a questionnaire for care taker.
  The Neuropsychiatric Inventory (NPI) was developed to provide a means of assessing neuropsychiatric symptoms and psychopathology of patients with Alzheimer's disease and other neurodegenerative disorders (Cummings 1997). Ten behavioral and two neurovegetative areas are included in the NPI.
  The NPI is based on responses from an informed caregiver, preferably one living with the patient. A caregiver can be defined as a person spending at least 4 hours per day at least 4 days per week with the patient and who is knowledgeable about the patient's daytime and nighttime behaviors.
  The total NPI score is the sum of all items. It varies from 0 to 120 for the behavioral domains and from 0 to 144 for all 12 domains.
Neuropsychiatric Inventory (NPI) (Care Taker) | month 1
  The NPI stands for "Neuropsychiatric Inventory". It is a questionnaire for care taker.
  The Neuropsychiatric Inventory (NPI) was developed to provide a means of assessing neuropsychiatric symptoms and psychopathology of patients with Alzheimer's disease and other neurodegenerative disorders (Cummings 1997). Ten behavioral and two neurovegetative areas are included in the NPI.
  The NPI is based on responses from an informed caregiver, preferably one living with the patient. A caregiver can be defined as a person spending at least 4 hours per day at least 4 days per week with the patient and who is knowledgeable about the patient's daytime and nighttime behaviors.
  The total NPI score is the sum of all items. It varies from 0 to 120 for the behavioral domains and from 0 to 144 for all 12 domains.
Neuropsychiatric Inventory (NPI) (Care Taker) | month 3
  The NPI stands for "Neuropsychiatric Inventory". It is a questionnaire for care taker.
  The Neuropsychiatric Inventory (NPI) was developed to provide a means of assessing neuropsychiatric symptoms and psychopathology of patients with Alzheimer's disease and other neurodegenerative disorders (Cummings 1997). Ten behavioral and two neurovegetative areas are included in the NPI.
  The NPI is based on responses from an informed caregiver, preferably one living with the patient. A caregiver can be defined as a person spending at least 4 hours per day at least 4 days per week with the patient and who is knowledgeable about the patient's daytime and nighttime behaviors.
  The total NPI score is the sum of all items. It varies from 0 to 120 for the behavioral domains and from 0 to 144 for all 12 domains.
IADL (Care Taker) | immediately post-treatment
  Questionnaire for care taker. IADL stands for "Instrumental Activities of Daily Living". Lawton's Instrumental Activities of Daily Living Scale (IADL) is an instrument to assess independent living skills (Lawton 1969). This questionnaire is supposed to be completed by the patient as well as by a person familiar with the patient. There are 8 domains of function measured with the Lawton IADL scale: Telephone, Shopping, Food preparation, Housekeeping, Laundry, Mode of transportation, Medication, Finances.
  The Total Score is a sum of all domains. The total score ranges from 0 (low function, dependent) to 8 (high function, independent). For male patients the highest possible score is 5 (due to expected zero scores for food preparation, housekeeping, and laundry).
IADL (Care Taker) | month 1
  Questionnaire for care taker. IADL stands for "Instrumental Activities of Daily Living". Lawton's Instrumental Activities of Daily Living Scale (IADL) is an instrument to assess independent living skills (Lawton 1969). This questionnaire is supposed to be completed by the patient as well as by a person familiar with the patient. There are 8 domains of function measured with the Lawton IADL scale: Telephone, Shopping, Food preparation, Housekeeping, Laundry, Mode of transportation, Medication, Finances.
  The Total Score is a sum of all domains. The total score ranges from 0 (low function, dependent) to 8 (high function, independent). For male patients the highest possible score is 5 (due to expected zero scores for food preparation, housekeeping, and laundry).
IADL (Care Taker) | month 3
  Questionnaire for care taker. IADL stands for "Instrumental Activities of Daily Living". Lawton's Instrumental Activities of Daily Living Scale (IADL) is an instrument to assess independent living skills (Lawton 1969). This questionnaire is supposed to be completed by the patient as well as by a person familiar with the patient. There are 8 domains of function measured with the Lawton IADL scale: Telephone, Shopping, Food preparation, Housekeeping, Laundry, Mode of transportation, Medication, Finances.
  The Total Score is a sum of all domains. The total score ranges from 0 (low function, dependent) to 8 (high function, independent). For male patients the highest possible score is 5 (due to expected zero scores for food preparation, housekeeping, and laundry).
Bayer Activities of Daily Living Scale (B-ADL) | [ Time Frame: immediately post-treatment ]
  The B-ADL scale is used to assess deficits in the performance of everyday activities. The scale's main target group is community dwelling patients who suffer from mild cognitive impairment or mild-to-moderate dementia. It comprises 25 items. Each item is scored from 1 (no difficulties at all) to 10 (always difficulties). The global B-ADL score is the arithmetic mean of all items.
Bayer Activities of Daily Living Scale (B-ADL) | [ Time Frame: month 1 ]
  The B-ADL scale is used to assess deficits in the performance of everyday activities. The scale's main target group is community dwelling patients who suffer from mild cognitive impairment or mild-to-moderate dementia. It comprises 25 items. Each item is scored from 1 (no difficulties at all) to 10 (always difficulties). The global B-ADL score is the arithmetic mean of all items.
Bayer Activities of Daily Living Scale (B-ADL) | [ Time Frame: month 3 ]
  The B-ADL scale is used to assess deficits in the performance of everyday activities. The scale's main target group is community dwelling patients who suffer from mild cognitive impairment or mild-to-moderate dementia. It comprises 25 items. Each item is scored from 1 (no difficulties at all) to 10 (always difficulties). The global B-ADL score is the arithmetic mean of all items.
Geriatric Depression Scale - short form (GDS-15) | [ Time Frame: immediately post-treatment ]
  The Geriatric Depression Scale (GDS) is a questionnaire to assess depression in the elderly population. This scale generates self-evaluation scores concerning various aspects with relevance for the depressive disease (e.g. mood, drive, anxiety). The short form contains 15 items. The GDS-15 score ranges from 0 (normal state) to 15 (severe depression).
Geriatric Depression Scale - short form (GDS-15) | [ Time Frame: month 1 ]
  The Geriatric Depression Scale (GDS) is a questionnaire to assess depression in the elderly population. This scale generates self-evaluation scores concerning various aspects with relevance for the depressive disease (e.g. mood, drive, anxiety). The short form contains 15 items. The GDS-15 score ranges from 0 (normal state) to 15 (severe depression).
Geriatric Depression Scale - short form (GDS-15) | [ Time Frame: month 3 ]
  The Geriatric Depression Scale (GDS) is a questionnaire to assess depression in the elderly population. This scale generates self-evaluation scores concerning various aspects with relevance for the depressive disease (e.g. mood, drive, anxiety). The short form contains 15 items. The GDS-15 score ranges from 0 (normal state) to 15 (severe depression).
Leisure Behavior (FZV; German: Freizeitverhalten) | [ Time Frame: immediately post-treatment ]
  The leisure behavior questionnaire has 25 items covering the following activities: information / entertainment, active movement, social interactions, creative activities, church / cultural / educational activities. The frequency of each activity is rated on a Likert-Scale from 0 (never) to 6 (daily). The total score (0-6) is calculated as the average of all 25 items.
Leisure Behavior (FZV; German: Freizeitverhalten) | [ Time Frame: month 1 ]
  The leisure behavior questionnaire has 25 items covering the following activities: information / entertainment, active movement, social interactions, creative activities, church / cultural / educational activities. The frequency of each activity is rated on a Likert-Scale from 0 (never) to 6 (daily). The total score (0-6) is calculated as the average of all 25 items.
Leisure Behavior (FZV; German: Freizeitverhalten) | [ Time Frame: month 3 ]
  The leisure behavior questionnaire has 25 items covering the following activities: information / entertainment, active movement, social interactions, creative activities, church / cultural / educational activities. The frequency of each activity is rated on a Likert-Scale from 0 (never) to 6 (daily). The total score (0-6) is calculated as the average of all 25 items.
anatomical Magnetic Resonance Imaging (MRI) | immediately post-treatment
  3 Tesla Magnetic Resonance Imaging (MRI) for safety reasons: no bleeding or anatomical changes to the brain.
functional Magnetic Resonance Imaging (fMRI) | immediately post-treatment
  3 Tesla functional Magnetic Resonance Imaging (MRI) to analyze brain activation and connectivity after TPS. This will be done according to Sperling 2001.

CONTACTS AND LOCATIONS:
Overall Officials: Roland Beisteiner, Prof., Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Background] Chandler MJ, Lacritz LH, Hynan LS, Barnard HD, Allen G, Deschner M, Weiner MF, Cullum CM. A total score for the CERAD neuropsychological battery. Neurology. 2005 Jul 12;65(1):102-6. doi: 10.1212/01.wnl.0000167607.63000.38. PMID 16009893
- [Background] Fillenbaum GG, van Belle G, Morris JC, Mohs RC, Mirra SS, Davis PC, Tariot PN, Silverman JM, Clark CM, Welsh-Bohmer KA, Heyman A. Consortium to Establish a Registry for Alzheimer's Disease (CERAD): the first twenty years. Alzheimers Dement. 2008 Mar;4(2):96-109. doi: 10.1016/j.jalz.2007.08.005. PMID 18631955
- [Background] Hallikainen I, Hanninen T, Fraunberg M, Hongisto K, Valimaki T, Hiltunen A, Karppi P, Sivenius J, Soininen H, Koivisto AM; ALSOVA study group. Progression of Alzheimer's disease during a three-year follow-up using the CERAD-NB total score: Kuopio ALSOVA study. Int Psychogeriatr. 2013 Aug;25(8):1335-44. doi: 10.1017/S1041610213000653. Epub 2013 May 16. PMID 23676340
- [Background] Rosen WG, Mohs RC, Davis KL. A new rating scale for Alzheimer's disease. Am J Psychiatry. 1984 Nov;141(11):1356-64. doi: 10.1176/ajp.141.11.1356. PMID 6496779
- [Background] Morris JC, Mohs RC, Rogers H, Fillenbaum G, Heyman A. Consortium to establish a registry for Alzheimer's disease (CERAD) clinical and neuropsychological assessment of Alzheimer's disease. Psychopharmacol Bull. 1988;24(4):641-52. No abstract available. PMID 3249766
- [Background] Ehrensperger MM, Berres M, Taylor KI, Monsch AU. Early detection of Alzheimer's disease with a total score of the German CERAD. J Int Neuropsychol Soc. 2010 Sep;16(5):910-20. doi: 10.1017/S1355617710000822. Epub 2010 Aug 4. PMID 20682088
- [Background] Rossetti HC, Munro Cullum C, Hynan LS, Lacritz LH. The CERAD Neuropsychologic Battery Total Score and the progression of Alzheimer disease. Alzheimer Dis Assoc Disord. 2010 Apr-Jun;24(2):138-42. doi: 10.1097/WAD.0b013e3181b76415. PMID 20505431
- [Background] Seo EH, Lee DY, Lee JH, Choo IH, Kim JW, Kim SG, Park SY, Shin JH, Do YJ, Yoon JC, Jhoo JH, Kim KW, Woo JI. Total scores of the CERAD neuropsychological assessment battery: validation for mild cognitive impairment and dementia patients with diverse etiologies. Am J Geriatr Psychiatry. 2010 Sep;18(9):801-9. doi: 10.1097/JGP.0b013e3181cab764. PMID 20220577
- [Background] Irizarry MC, Webb DJ, Bains C, Barrett SJ, Lai RY, Laroche JP, Hosford D, Maher-Edwards G, Weil JG. Predictors of placebo group decline in the Alzheimer's disease Assessment Scale-cognitive subscale (ADAS-Cog) in 24 week clinical trials of Alzheimer's disease. J Alzheimers Dis. 2008 Jul;14(3):301-11. doi: 10.3233/jad-2008-14304. PMID 18599956
- [Background] Robert P, Ferris S, Gauthier S, Ihl R, Winblad B, Tennigkeit F. Review of Alzheimer's disease scales: is there a need for a new multi-domain scale for therapy evaluation in medical practice? Alzheimers Res Ther. 2010 Aug 26;2(4):24. doi: 10.1186/alzrt48. PMID 20796301
- [Background] Lehrner, J.; Maly, J.; Gleiß, A.; Auff, E. & Dal-Bianco, P., Demenzdiagnostik mit Hilfe der Vienna Neuropsychologischen Testbatterie (VNTB): Standardisierung, Normierung und Validierung, Psychol. Österreich, 4, 358-365, 2007.
- [Background] Shulman, K. I.; Shedletsky, R. & Silver, I. L.The challenge of time: Clock-drawing and cognitive function in the elderly. International journal of geriatric psychiatry, Wiley Online Library 1: 135-140, 1986.
- [Background] Kogler, B. Subjective Memory Complaint in Mild Cognitive Impairment, Alzheimer's Disease and Parkinson's Disease. Vienna: University of Vienna, 2013
- [Background] Lehrner J, Moser D, Klug S, Gleiss A, Auff E, Dal-Bianco P, Pusswald G. Subjective memory complaints, depressive symptoms and cognition in patients attending a memory outpatient clinic. Int Psychogeriatr. 2014 Mar;26(3):463-73. doi: 10.1017/S1041610213002263. Epub 2013 Dec 5. PMID 24308705
- [Background] Lawton MP, Brody EM. Assessment of older people: self-maintaining and instrumental activities of daily living. Gerontologist. 1969 Autumn;9(3):179-86. No abstract available. PMID 5349366
- [Background] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369
- [Background] Shah P, Gaule A, Sowden S, Bird G, Cook R. The 20-item prosopagnosia index (PI20): a self-report instrument for identifying developmental prosopagnosia. R Soc Open Sci. 2015 Jun 24;2(6):140343. doi: 10.1098/rsos.140343. eCollection 2015 Jun. PMID 26543567
- [Background] Cummings JL. The Neuropsychiatric Inventory: assessing psychopathology in dementia patients. Neurology. 1997 May;48(5 Suppl 6):S10-6. doi: 10.1212/wnl.48.5_suppl_6.10s. PMID 9153155
- [Background] Sperling RA, Bates JF, Cocchiarella AJ, Schacter DL, Rosen BR, Albert MS. Encoding novel face-name associations: a functional MRI study. Hum Brain Mapp. 2001 Nov;14(3):129-39. doi: 10.1002/hbm.1047. PMID 11559958
- [Derived] Matt E, Mitterwallner M, Radjenovic S, Grigoryeva D, Weber A, Stogmann E, Domitner A, Zettl A, Osou S, Beisteiner R. Ultrasound Neuromodulation With Transcranial Pulse Stimulation in Alzheimer Disease: A Randomized Clinical Trial. JAMA Netw Open. 2025 Feb 3;8(2):e2459170. doi: 10.1001/jamanetworkopen.2024.59170. PMID 40009384